CLINICAL TRIAL: NCT03786302
Title: Comparison of the Regenerative Ability of Tailored Amorphous Multiporous Bioglass and Biodentine in Pulpotomized Primary Teeth
Brief Title: Regenerative Ability of TAMP BG and BD in Pulpotomized Primary Teeth
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Failure rate was 100% in one arm of the study (the intervention)
Sponsor: Nourhan M.Aly (Other)
Collaborators: Alexandria University (Other)
Responsible Party: Sponsor-Investigator, Nourhan M.Aly, Clinical Instructor, University of Alexandria
Organization: University of Alexandria (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Bioglass in pulpotomized teeth
Record Dates: First submitted 2018-12-18; First posted 2018-12-26 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Pulpotomy
Keywords: TAMP BG; Biodentine; Regenerative materials; pulp therapy
MeSH Terms: interventions — tricalcium silicate

STUDY DESIGN:
Intervention Model Description: Study group (assigned to TAMP bioglass), and Control group (assigned to Biodentine ™).
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The operator will not be blinded to the treatment type. However, the participants, their care givers, the expert assessing the histologic and inflammatory changes and the statistician will be blinded to the treatment groups.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAMP bioglass (Experimental): Tailored amorphous multiporous bioglass (TAMP-BG) of 70% SiO2 / 30% CaO was prepared according to Wang et al. (2011, 2013) in the tissue engineering lab, Faculty of Dentistry, Alexandria University as follows: Scaffolds were grounded to 180- to 300-μm particle size and sterilized at 180°C for 2 hours. The resulting powder was mixed with distilled water to obtain a putty like consistency that was carried to the pulp chamber and condensed lightly on the pulp stumps.
  Interventions: Drug: TAMP bioglass
- Biodentine ™ (Active Comparator): Biodentine ™ (BD) pre-dosed capsule were gently tapped on a hard surface to diffuse the powder. Five drops of the liquid from the single dose dispenser were poured into the capsule and mixed for 30 seconds at 4,200 rpm in an amalgamator according to manufacturer's instructions to obtain putty- like consistency. (Powder-liquid system). It was then be carried to the pulp chamber and condensed lightly on the pulp stumps. Final restoration was applied after 12 minutes, allowing Biodentine ™ to set.
  Interventions: Drug: Biodentine

INTERVENTIONS:
Drug: TAMP bioglass — TAMP bioglass compared to Biodentine in the regeneration on pulpotomized primary teeth
  Other Names: 70S30C bioglass
  Arms: TAMP bioglass
Drug: Biodentine — TAMP bioglass compared to Biodentine in the regeneration on pulpotomized primary teeth
  Arms: Biodentine ™

SUMMARY:
The aim of this study was to assess clinically, radiographically, and histologically the regenerative ability of Tailored Amorphous Mulioporous (TAMP-BG) bioglass in comparison to Biodentine™ (BD) in pulpotomized primary teeth.

DETAILED DESCRIPTION:
The study was a parallel design, randomized controlled clinical trial It was conducted in the out-patient clinic of the Pediatric Dentistry and Dental public health department after obtaining the guardians consent. The sample size was calculated to be 35 teeth per group. The teeth were randomly and equally assigned to either BD or TAMP-BG groups.The treatment follow-up was scheduled at 1, 3, 6, 9 and 12 months. The study was terminated for ethical considerations after showing significant clinical failure in the TAMP-BG group and after performing interim analysis.

ELIGIBILITY:
Inclusion Criteria:

* Children free of any systemic disease or special health care needs.
* Children not receiving any anti-inflammatory medication.
* Cooperative children (positive/ definitely positive) according to Frankl's behavior rating scale.
* Restorable teeth.
* Teeth with vital carious pulp exposure that will bleed upon entering the pulp chamber and not requiring more than 5 minutes to achieve hemostasis after coronal pulp amputation.
* Teeth indicated for extraction for orthodontic purposes with the previously mentioned criteria (required for a subgroup for assessment of histological and inflammatory response outcomes).

Exclusion Criteria:

* Teeth with clinical or radiographic signs of pulp degeneration.

Ages: 5 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 102 (Actual)
Dates: Start 2016-12-06 (Actual); Primary Completion 2018-08-15 (Actual); Study Completion 2018-10-20 (Actual)

PRIMARY OUTCOMES:
Absence of clinical signs of pulp degeneration. | 1 month postoperatively
  Teeth were considered clinically successful when they showed no signs of pain, sensitivity to percussion, swelling, fistula or pathologic mobility
Percentage of Teeth with no clinical signs of pulp degeneration. | 3 months postoperatively
  Teeth were considered clinically successful when they showed no signs of pain, sensitivity to percussion, swelling, fistula or pathologic mobility
Percentage of Teeth with no clinical signs of pulp degeneration. | 6 months postoperatively
  Teeth were considered clinically successful when they showed no signs of pain, sensitivity to percussion, swelling, fistula or pathologic mobility
Percentage of Teeth with no clinical signs of pulp degeneration. | 9 months postoperatively
  Teeth were considered clinically successful when they showed no signs of pain, sensitivity to percussion, swelling, fistula or pathologic mobility
Percentage of Teeth with no clinical signs of pulp degeneration. | 12 months postoperatively
  Teeth were considered clinically successful when they showed no signs of pain, sensitivity to percussion, swelling, fistula or pathologic mobility
Percentage of Teeth with no radiographic signs of pulp degeneration. | 6 months postoperatively
  Digital postoperative periapical radiographs were obtained and assessed for signs of pulp degeneration. Teeth were considered radiographically successful when they showed no periapical or interradicular radiolucency, abnormal root resorption or periodontal ligament space widening
Percentage of Teeth with no radiographic signs of pulp degeneration. | 12 months postoperatively
  Digital postoperative periapical radiographs were obtained and assessed for signs of pulp degeneration. Teeth were considered radiographically successful when they showed no periapical or interradicular radiolucency, abnormal root resorption or periodontal ligament space widening

SECONDARY OUTCOMES:
Percentage of teeth with radiographic evidence of dentin bridge formation | 6 months postoperatively
  Assessed using digital radiographs
Percentage of teeth with radiographic evidence of dentin bridge formation | 12 months postoperatively
  Assessed using digital radiographs
Dentin bridge formation using light microscopy | 6 weeks
  After tooth extraction, histological assessment will be done according to Horsted et al's (1981) and Shayegan et al's (2012) modified criteria.
  0= No hard tissue formation.
  1. Incomplete hard tissue formation.
  2. Thick hard tissue formation.
Inflammatory response using light microscopy | 6 weeks
  After tooth extraction, histological assessment will be done according to Horsted et al's (1981) and Shayegan et al's (2012) modified criteria. A. Inflammatory cell response:
  0= None or a few scattered inflammatory cells beneath the site of pulp exposure.
  1. Mild inflammatory cells (either acute or chronic).
  2. Moderate inflammatory cell infiltration involving the cervical third of radicular pulp.
  3. Severe inflammatory cell infiltration involving the coronal third of radicular pulp.
  B. Tissue disorganization:
  0= Normal tissue beneath the site of pulp exposure.
  1. Odontoblast-like cells, odontoblasts, and pulp tissue pattern disorganization.
  2. General disorganization of the pulp tissue pattern.
  3. Pulp necrosis.
The Enzyme-Linked Immunosorbent Assay (ELISA) analysis. | 6 weeks
  After extraction, the tooth will be sectioned under copious water cooling and all remaining pulp tissue will be harvested gently from the radicular portion and stored until the time of assaying. For the ELISA assaying, the frozen pulp samples will be thawed for 15 minutes, and crushed with a glass rod in the eppendorf tube to elute the cytokines from the pulp tissue. IL-8 and IL-10 will be measured using ElISA Kits according to the instructions supplied with the kit and the ratio of IL-8/IL-10 will be taken as an indicator of pulpal inflammation. Cytokines' concentration will be calculated according to the weight of the pulp tissue.

CONTACTS AND LOCATIONS:
Overall Officials: Yasmine I El-Hamouly, MSc, Principal Investigator — Alexandria University; Karin ML Dowidar, PhD, Study Director — Alexandria University; Samia Soliman, PhD, Study Director — Alexandria University; Dalia AM Talaat, PhD, Study Director — Alexandria University; Rania M El Backly, PhD, Study Director — Alexandria University
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt

REFERENCES:
- [Background] Wang S, Falk MM, Rashad A, Saad MM, Marques AC, Almeida RM, Marei MK, Jain H. Evaluation of 3D nano-macro porous bioactive glass scaffold for hard tissue engineering. J Mater Sci Mater Med. 2011 May;22(5):1195-203. doi: 10.1007/s10856-011-4297-4. Epub 2011 Mar 29. PMID 21445655
- [Background] Wang S, Kowal TJ, Marei MK, Falk MM, Jain H. Nanoporosity significantly enhances the biological performance of engineered glass tissue scaffolds. Tissue Eng Part A. 2013 Jul;19(13-14):1632-40. doi: 10.1089/ten.TEA.2012.0585. Epub 2013 Mar 26. PMID 23427819
- [Background] Stanley HR, Clark AE, Pameijer CH, Louw NP. Pulp capping with a modified bioglass formula (#A68-modified). Am J Dent. 2001 Aug;14(4):227-32. PMID 11699742
- [Background] Horsted P, El Attar K, Langeland K. Capping of monkey pulps with Dycal and a Ca-eugenol cement. Oral Surg Oral Med Oral Pathol. 1981 Nov;52(5):531-53. doi: 10.1016/0030-4220(81)90366-2. PMID 6946381
- [Background] Shayegan A, Jurysta C, Atash R, Petein M, Abbeele AV. Biodentine used as a pulp-capping agent in primary pig teeth. Pediatr Dent. 2012 Nov-Dec;34(7):e202-8. PMID 23265156
- [Derived] Elhamouly Y, El Backly RM, Talaat DM, Omar SS, El Tantawi M, Dowidar KML. Tailored 70S30C Bioactive glass induces severe inflammation as pulpotomy agent in primary teeth: an interim analysis of a randomised controlled trial. Clin Oral Investig. 2021 Jun;25(6):3775-3787. doi: 10.1007/s00784-020-03707-5. Epub 2021 Jan 6. PMID 33409691